CLINICAL TRIAL: NCT04958915
Title: Application Value of Flexion Position MRI in Diagnosis of Anterior Cruciate Ligament Injury and Patellofemoral Instability
Brief Title: Application of FMRI in Diagnosis of Anterior Cruciate Ligament Injury
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018014
Record Dates: First submitted 2021-06-28; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2018-03

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 30 ° flexion position: Scan the knee at 30° flexion
  Interventions: Diagnostic Test: Knee joint 30° flexion scan
- conventional flexion position: Routine body scan of the knee joint

INTERVENTIONS:
Diagnostic Test: Knee joint 30° flexion scan — The patient was placed in the supine position, and the knee joint was naturally placed in the knee joint special coil, and the knee joint 30° flexion position scan.
  Groups: 30 ° flexion position

SUMMARY:
1. To compare the knee joint MRI 30 ° The flexion position was similar to that of conventional knee joint coil (about 17 °） The advantages and disadvantages in the description and diagnosis of anterior cruciate ligament injury;,2. To compare the knee joint MRI 30 ° The flexion position was similar to that of conventional knee joint coil (about 17 °） Advantages and disadvantages in description and diagnosis of patellofemoral instability

DETAILED DESCRIPTION:
Magnetic resonance imaging is widely used in the imaging diagnosis of knee joint injury. At present, there are two kinds of scanning coils used in our country. One is flexible surface coil, and the patient is 0 ° Scan in the straight position. The other is the special coil for the knee joint. At this time, because the coil itself is hard material and has a certain height, the patient is actually in the knee joint micro bending position (about 17 ° 1) Scan. However, it may not be accurate enough to evaluate ACL injury and patellofemoral instability with knee scan in extension and micro flexion position.,1、 Previous literatures have shown that flexion position is superior to extension position in the description and diagnosis of anterior cruciate ligament injury. The main reasons include: ① in extension position, the femoral attachment is wider and flat, with the increase of flexion angle, the anterior cruciate ligament fiber bundle is twisted, and the femoral segment is narrower in sagittal position, Thus, it can be clearly shown as a cylindrical bundle structure 2; ② The normal ACL was tensioned in the extension position, so the femoral attachment area was not well displayed. With the increase of flexion angle, the femoral segment separated from the intercondylar crest area, and the volume of intercondylar fossa increased; ③ Due to the influence of partial volume artifacts in the extension position, the normal anterior cruciate ligament may also show uneven MRI signal, which is similar to injury, resulting in false positive, while the flexion position can reduce partial volume artifacts. However, there are few studies on the advantages and disadvantages of flexion and micro flexion scanning in the description and diagnosis of anterior cruciate ligament injury at home and abroad.,2、 The medical research of patellofemoral instability found that in the early stage of knee flexion, the patella of normal people began to move to the medial side of the knee while sliding from the starting position to the distal side ° The patella moved inward gradually to the maximum, then turned to the lateral and moved to the knee flexion of 40 ° The patella returned to the median line 4. The patients with patellofemoral instability were 15 °- forty-five ° The center of patella moved from the initial position to the lateral position continuously for 5, so 30 ° The difference between normal people and patients may be more significant.,The purpose of this study is to explore 30 cases ° Application value of flexion position in diagnosis of anterior cruciate ligament injury and patellofemoral instability.

2.Image analysis：Comparison of the diagnosis of anterior cruciate ligament injury between conventional scan position and 30°flexion scan

(1) Two radiologists respectively evaluated the injury of the anterior cruciate ligament.

The evaluation criteria for the full length display status are as follows: 3 points: The anterior cruciate ligament is continuously displayed on multiple levels or the full length is displayed in one level, without obvious artifacts; 2 points: The full length of the anterior cruciate ligament cannot be displayed completely but the section can be displayed, there are artifacts but it does not affect the observation; (1)point: The full length of the anterior cruciate ligament cannot be identified or artifacts affect the observation. The evaluation criteria for the display status of the tearing point and stump are as follows: (3) points: The tear point and stump of the ACL are clearly displayed (2) points: One of the torn points or stumps of the ACL can be clearly displayed, and the other cannot be clearly displayed (1) point: The tear point and stump of the ACL cannot be clearly displayed

ELIGIBILITY:
Inclusion Criteria: Hospitalized patients who have a clear history of knee joint sports injury who are planning to undergo knee arthroscopy -

Exclusion Criteria: MR examination found to have the following diseases: rheumatoid arthritis, septic arthritis, tumor, joint fibrosis; History of knee surgery.

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients or inpatients who were clinically diagnosed with patellofemoral instability and planned to undergo knee MRI examination from March 2018 to October 2018
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-10-13 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Damage diagnosis | 2019.1.15-2019.1.30
  Arthroscopy was used as the gold standard to evaluate the ACCURACY of the two methods in the diagnosis of ligament injury

CONTACTS AND LOCATIONS:
Overall Officials: Huishu Yuan, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No